CLINICAL TRIAL: NCT02968888
Title: Effects of Whey and Casein Supplementation on Acute Anabolic Responses in Muscle After Strength Training in Young and Elderly
Brief Title: Anabolic Effects of Whey and Casein After Strength Training in Young and Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: Tine (Industry); The Research Council of Norway (Other); Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Havard Hamarsland, PhD student, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Tine acute
Record Dates: First submitted 2016-11-10; First posted 2016-11-21 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Healthy; Young; Elderly
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Milk (Placebo Comparator): Participants performed a bout of strength training and consumed 20g of milk protein
  Interventions: Other: Strength training; Dietary Supplement: Milk 1%
- Whey protein concentrate 80 (Experimental): Participants performed a bout of strength training and consumed 20g of whey protein concentrate 80
  Interventions: Other: Strength training; Dietary Supplement: Whey protein concentrate 80
- Native whey (Experimental): Participants performed a bout of strength training and consumed 20g of native whey
  Interventions: Other: Strength training; Dietary Supplement: Native whey

INTERVENTIONS:
Other: Strength training
Dietary Supplement: Milk 1%
  Arms: Milk
Dietary Supplement: Whey protein concentrate 80
  Arms: Whey protein concentrate 80
Dietary Supplement: Native whey
  Arms: Native whey

SUMMARY:
The aim of this study is to investigate the acute anabolic effects of native whey, whey protein concentrate 80 (WPC-80) and milk after a bout of strength training in young and elderly. The investigators hypothesize that native whey will give a greater stimulation of muscle protein synthesis and intracellular anabolic signaling than WPC-80, and that WPC-80 will give a stronger stimulus than milk.

DETAILED DESCRIPTION:
Increasing or maintaining muscle mass is of great importance for populations ranging from athletes to patients and elderly. Resistance exercise and protein ingestion are two of the most potent stimulators of muscle protein synthesis. Both the physical characteristic of proteins (e.g. different digestion rates of whey and casein) and the amino acid composition, affects the potential of a certain protein to stimulate muscle protein synthesis. Given its superior ability to rapidly increase blood leucine concentrations to high levels, whey is often considered the most potent protein source to stimulate muscle protein synthesis. Native whey protein is produced by filtration of unprocessed milk. Consequently, native whey has different characteristics than WPC-80, which is exposed to heating and acidification. Because of the direct filtration of unprocessed milk, native whey is a more intact protein compared with WPC-80. Of special interest is the higher amounts of the highly anabolic amino acid leucine in native whey.

The higher levels of leucine can be of great interest for elderly individuals as some studies in elderly has shown an anabolic resistance to the effects of protein feeding and strength training. By increasing levels of leucine one might overcome this anabolic resistance in the elderly.

The aim of this double-blinded, randomized, partial cross-over study is to compare the acute fractional protein synthesis and intracellular signaling response to a bout of strength training and intake of 20 grams of protein from either native whey, whey protein concentrate 80 or milk, in young and old individuals. Furthermore, the investigators wil investigate fractional protein breakdown, markers of protein breakdown, amino acid concentrations in blood.

The investigators hypothesize that native whey will induce a greater anabolic response than whey protein concentrate 80, and that whey protein concentrate 80 will give a stronger anabolic response than milk.

ELIGIBILITY:
Inclusion Criteria:

* Healthy in the sense that they can conduct training and testing
* Able to understand Norwegian language written and oral
* Between 18 and 45, or above 70 years of age

Exclusion Criteria:

* Diseases or injuries contraindicating participation
* Use of dietary supplements (e.g. proteins, vitamins and creatine)
* Lactose intolerance
* Allergy to milk
* Allergy towards local anesthetics (xylocain)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Mixed muscle fractional synthetic rate | Three to one hours prior to a bout of strength training and protein consumption
  A continous infusion of a stable isotope (phe D5) is used to measure incorporation of tracer into muscle (biopsies from m. vastus lateralis)
Mixed muscle fractional synthetic rate | One to five hours after a bout of strength training and protein consumption
  A continous infusion of a stable isotope (phe D5) is used to measure incorporation of tracer into muscle (biopsies from m. vastus lateralis)
Mixed muscle fractional synthetic rate | From three to five hours after a bout of strength training and protein consumption
  Two boluses of tracer (phe13C6 and phe15N) was used to measure incorporation of tracer into muscle (biopsies from m. vastus lateralis)
Mixed muscle fractional breakdown rate | From three to five hours after a bout of strength training and protein consumption
  Two boluses of tracer (phe13C6 and phe15N) was used to measure the dilution of tracer in muscle (biopsies from m. vastus lateralis)

SECONDARY OUTCOMES:
Ratio of phosphorylated to total ribosomal protein S6 kinase beta-1(P70S6K) change from baseline | 30 min before, 1, 2.5 and 5 hours after training and protein intake
  Biopsies from m. Vastus Lateralis was analyzed by western blot
Phosphorylation of phosphorylated to total eukaryotic elongation factor 2 (eEF-2) change from baseline | 30 min before, 1, 2.5 and 5 hours after training and protein intake
  Biopsies from m. Vastus Lateralis was analyzed by western blot
Phosphorylation of phosphorylated to total eukaryotic translation initiation factor 4E-binding protein 1 (4EBP-1) change from baseline | 30 min before, 1, 2.5 and 5 hours after training and protein intake
  Biopsies from m. Vastus Lateralis was analyzed by western blot
Intracellular translocation of forkhead box O3 (FOXO3a) change from baseline | 30 min before, 1, 2.5 and 5 hours after training and protein intake
  Biopsies from m. Vastus Lateralis was analyzed by western blot
Intracellular translocation of muscle RING-finger protein-1 (Murf-1) change from baseline | 30 min before, 1, 2.5 and 5 hours after training and protein intake
  Biopsies from m. Vastus Lateralis was analyzed by western blot
Intracellular translocation of Atrogin1 change from baseline | 30 min before, 1, 2.5 and 5 hours after training and protein intake
  Biopsies from m. Vastus Lateralis was analyzed by western blot
Ubiquitin | 30 min before, 1, 2.5 and 5 hours after training and protein intake
  Biopsies from m. Vastus Lateralis was analyzed by western blot
Plasma amino acid concentration | 180 and 60 min before, and 45, 60, 75, 120, 160, 180, 200, 220 and 300 min after training and protein intake
Muscle force generating capacity change from baseline | 15 min before, 15 and 300 min after, and 24 hours after training and protein intake
  Measured as unilateral isometric knee extension force (Nm) with 90° in the hip and knee joints.
Plasma glucose | 180 and 60 min before, and 45, 60, 75, 120, 160, 180, 200, 220 and 300 min after training and protein intake
Plasma insulin | 180 and 60 min before, and 45, 60, 75, 120, 160, 180, 200, 220 and 300 min after training and protein intake
Serum urea | 180 and 60 min before, and 60, 10, 180 and 300 min after training and protein intake
Serum ureic acid | 180 and 60 min before, and 60, 10, 180 and 300 min after training and protein intake
Serum creatine kinase | 180 and 60 min before, and 60, 10, 180 and 300 min after training and protein intake
Change in ATP-binding cassette transporter (ABCA1) messenger ribonucleic acid (mRNA) | 1 hour after training and protein intake
Change in ABCA1 mRNA | 5 hous after training and protein intake
Change in BRCA1-A complex subunit Abraxas (ABRA1) mRNA | 1 hour after training and protein intake
Change in ABRA1 mRNA | 5 hours after training and protein intake
Change in alfa-actin (ACTA1) mRNA | 1 hour after training and protein intake
Change in ACTA1 mRNA | 5 hours after training and protein intake
Change in C-C motif chemokine 2 (CCL2) mRNA | 1 hour after training and protein intake
Change in CCL2 mRNA | 5 hours after training and protein intake
Change in C-C motif chemokine 3 (CCL3) mRNA | 1 hour after training and protein intake
Change in CCL3 mRNA | 5 hours after training and protein intake
Change in C-C motif chemokine 5 (CCL5) mRNA | 1 hour after training and protein intake
Change in CCL5 mRNA | 5 hours after training and protein intake
Change in C-C motif chemokine 8 (CCL8) mRNA | 1 hour after training and protein intake
Change in CCL8 mRNA | 5 hours after training and protein intake
Change in platelet glycoprotein 4 (CD36) mRNA | 1 hour after training and protein intake
Change in CD36 mRNA | 5 hours after training and protein intake
Change in cholesterol 25-hydroxylase (CH25H) mRNA | 1 hour after training and protein intake
Change in CH25H mRNA | 5 hours after training and protein intake
Change in granulocyte colony-stimulating factor (CSF3) mRNA | 1 hour after training and protein intake
Change in CSF3 mRNA | 5 hours after training and protein intake
Change in C-X-C motif chemokine 16 (CXCL16) mRNA | 1 hour after training and protein intake
Change in CXCL16 mRNA | 5 hours after training and protein intake
Change in F-box only protein 32 (FBXO32) mRNA | 1 hour after training and protein intake
Change in FBXO32 mRNA | 5 hours after training and protein intake
Change in growth-regulated alpha protein (CXCL1) mRNA | 1 hour after training and protein intake
Change in CXCL1 mRNA | 5 hours after training and protein intake
Change in matrix metalloproteinase-9 (MMP9) mRNA | 1 hour after training and protein intake
Change in MMP9 mRNA | 5 hours after training and protein intake
Change in forkhead box protein O1 (FOXO1) mRNA | 1 hour after training and protein intake
Change in FOXO1 mRNA | 5 hours after training and protein intake
Change in forkhead box protein O3 (FOXO3A) mRNA | 1 hour after training and protein intake
Change in FOXO3A mRNA | 5 hours after training and protein intake
Change in hepatocyte growth factor (HGF) mRNA | 1 hour after training and protein intake
Change in HGF mRNA | 5 hours after training and protein intake
Change in insulin-like growth factor I (IGF1) mRNA | 1 hour after training and protein intake
Change in IGF1 mRNA | 5 hours after training and protein intake
Change in interleukin-10 (IL10) mRNA | 1 hour after training and protein intake
Change in IL10 mRNA | 5 hours after training and protein intake
Change in interleukin-17D (IL17D) mRNA | 1 hour after training and protein intake
Change in IL17D mRNA | 5 hours after training and protein intake
Change in interleukin-1B (IL1B) mRNA | 1 hour after training and protein intake
Change in IL1B mRNA | 5 hours after training and protein intake
Change in interleukin-1 receptor antagonist protein (IL1RN) mRNA | 1 hour after training and protein intake
Change in IL1RN mRNA | 5 hours after training and protein intake
Change in interleukin-6 (IL6) mRNA | 1 hour after training and protein intake
Change in IL6 mRNA | 5 hours after training and protein intake
Change in interleukin-8 (IL8) mRNA | 1 hour after training and protein intake
Change in IL8 mRNA | 5 hours after training and protein intake
Change in transcription factor jun-B (JUNB) mRNA | 1 hour after training and protein intake
Change in JUNB mRNA | 5 hours after training and protein intake
Change in kit ligand (KITLG) mRNA | 1 hour after training and protein intake
Change in KITLG mRNA | 5 hours after training and protein intake
Change in myostatin (MSTN) mRNA | 1 hour after training and protein intake
Change in MSTN mRNA | 5 hours after training and protein intake
Change in myosin-1 (MYH1) mRNA | 1 hour after training and protein intake
Change in MYH1 mRNA | 5 hours after training and protein intake
Change in myosin-2 (MYH2) mRNA | 1 hour after training and protein intake
Change in MYH2 mRNA | 5 hours after training and protein intake
Change in myosin-7 (MYH7) mRNA | 1 hour after training and protein intake
Change in MYH7 mRNA | 5 hours after training and protein intake
Change in oxysterols receptor LXR-alpha (NR1H3) mRNA | 1 hour after training and protein intake
Change in NR1H3 mRNA | 5 hours after training and protein intake
Change in nuclear receptor subfamily 4 group A member 3 (NR4A3) mRNA | 1 hour after training and protein intake
Change in NR4A3 mRNA | 5 hours after training and protein intake
Change in peroxisome proliferator-activated receptor gamma coactivator 1-alpha (PPARGC1A) mRNA | 1 hour after training and protein intake
Change in PPARGC1A mRNA | 5 hours after training and protein intake
Change in prostaglandin G/H synthase 2 (PTGS2) mRNA | 1 hour after training and protein intake
Change in PTGS2 mRNA | 5 hours after training and protein intake
Change in proton-coupled amino acid transporter 1 (SLC36A1) mRNA | 1 hour after training and protein intake
Change in SLC36A1 mRNA | 5 hours after training and protein intake
Change in sodium-coupled neutral amino acid transporter 2 (SLC38A2) mRNA | 1 hour after training and protein intake
Change in SLC38A2 mRNA | 5 hours after training and protein intake
Change in 4F2 cell-surface antigen heavy chain (SLC3A2) mRNA | 1 hour after training and protein intake
Change in SLC3A2 mRNA | 5 hours after training and protein intake
Change in large neutral amino acids transporter small subunit 1 (SLC7A5) mRNA | 1 hour after training and protein intake
Change in SLC7A5 mRNA | 5 hours after training and protein intake
Change in toll-like receptor 2 (TLR2) mRNA | 1 hour after training and protein intake
Change in TLR2 mRNA | 5 hours after training and protein intake
Change in tumor necrosis factor (TNF) mRNA | 1 hour after training and protein intake
Change in TNF mRNA | 5 hours after training and protein intake
Change in E3 ubiquitin-protein ligase TRIM63 (TRIM63) mRNA | 1 hour after training and protein intake
Change in E3 ubiquitin-protein ligase TRIM63 (TRIM63) mRNA | 5 hours after training and protein intake

CONTACTS AND LOCATIONS:
Locations (1):
- Norwegian School of Sport Sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hamarsland H, Nordengen AL, Nyvik Aas S, Holte K, Garthe I, Paulsen G, Cotter M, Borsheim E, Benestad HB, Raastad T. Native whey protein with high levels of leucine results in similar post-exercise muscular anabolic responses as regular whey protein: a randomized controlled trial. J Int Soc Sports Nutr. 2017 Nov 21;14:43. doi: 10.1186/s12970-017-0202-y. eCollection 2017. PMID 29200982